CLINICAL TRIAL: NCT00006230
Title: Open Label Phase II Study on RFS 2000 (9-Nitro-camptothecin, 9-NC) Administered as a "5 Days On-2 Days Off" Oral Treatment in Advanced Ovarian Cancer
Brief Title: Nitrocamptothecin in Treating Patients With Advanced Ovarian Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: EORTC-16996O; EORTC-16996O
Record Dates: First submitted 2000-09-11; First posted 2003-01-27 (Estimated); Last update posted 2012-09-24 (Estimated); Status verified 2012-09

CONDITIONS: Ovarian Cancer
Keywords: stage III ovarian epithelial cancer; stage IV ovarian epithelial cancer; recurrent ovarian epithelial cancer
MeSH Terms: conditions — Ovarian Neoplasms; Carcinoma, Ovarian Epithelial | interventions — rubitecan

INTERVENTIONS:
Drug: rubitecan

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of nitrocamptothecin in treating patients who have advanced ovarian cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the objective response rate and duration of response in patients with advanced ovarian cancer treated with nitrocamptothecin.
* Determine the probability of objective response as expressed by the response rate in patients treated with this regimen.
* Determine the toxicity of this regimen in these patients.

OUTLINE: This is a multicenter study. Patients are stratified according to disease status (sensitive vs refractory).

Patients receive oral nitrocamptothecin daily for 5 consecutive days each week for 3 weeks. Treatment continues every 3 weeks for a minimum of 2 courses in the absence of disease progression or unacceptable toxicity. Patients who achieve stable disease (SD) receive up to 4 additional courses past SD. Patients who achieve partial response (PR) or complete response (CR) receive a minimum of 2 additional courses past PR or CR.

Patients are followed every 6 weeks until disease progression or the initiation of another antitumor therapy.

PROJECTED ACCRUAL: A total of 28-50 patients (14-25 per stratum) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven metastatic or unresectable locally advanced progressive ovarian cancer that has failed first line platinum and taxane based regimen

  * Refractory disease defined by a relapse within 1 year after completion of first line therapy
  * Sensitive disease defined by a relapse greater than 1 year after completion of first line therapy
* Minimum of 1 target lesion that can be accurately measured in at least 1 dimension

  * At least 20 mm by conventional techniques OR
  * At least 10 mm by spiral CT scan
* No symptomatic brain metastases

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-2

Life expectancy:

* At least 3 months

Hematopoietic:

* Neutrophil count at least 2,000/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin less than 1.5 times upper limit of normal (ULN)
* Alkaline phosphatase, SGOT, and SGPT no greater than 2.5 times ULN (no greater than 5 times ULN if hepatic metastases present)

Renal:

* Creatinine no greater than 1.7 mg/dL

Cardiovascular:

* No ischemic heart disease within the past 6 months
* Normal 12 lead electrocardiogram

Other:

* Not pregnant or nursing
* Fertile patients must use effective contraception
* No unstable systemic disease or active uncontrolled infections
* No other prior or concurrent malignancy except adequately treated basal cell or squamous cell skin cancer or cone biopsied carcinoma of the cervix
* No psychological, familial, sociological, or geographical condition that would preclude compliance

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No concurrent filgrastim (G-CSF) with nitrocamptothecin

Chemotherapy:

* See Disease Characteristics
* Greater than 4 weeks since prior chemotherapy

Endocrine therapy:

* Not specified

Radiotherapy:

* Greater than 4 weeks since prior radiotherapy

Surgery:

* Greater than 2 weeks since prior major surgery

Other:

* No other concurrent anticancer agents
* No other concurrent investigational therapy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2000-05; Primary Completion 2003-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Fumoleau, MD, PhD, Study Chair — Centre Georges Francois Leclerc
Locations (13):
- Institut Jules Bordet, Brussels, Belgium
- France (5):
  - Centre Jean Perrin, Clermont-Ferrand
  - Centre de Lutte Contre le Cancer, Georges-Francois Leclerc, Dijon
  - CHU de la Timone, Marseille
  - CRLCC Nantes - Atlantique, Nantes-Saint Herblain
  - Centre Eugene Marquis, Rennes
- Rabin Medical Center - Beilinson Campus, Petah Tikva, Israel
- Azienda Ospedaliera di Padova, Padova (Padua), Italy
- Hospital Universitario 12 de Octubre, Madrid, Spain
- Switzerland (2):
  - Ospedale San Giovanni, Bellinzona
  - Clinique De Genolier, Genolier
- United Kingdom (2):
  - Newcastle General Hospital, Newcastle upon Tyne, England
  - Western General Hospital, Edinburgh, Scotland